CLINICAL TRIAL: NCT02169128
Title: Severe Soft Tissue Infections: Perspectives of Patients and Significant Others
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Karolinska Institutet (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SSTI
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Necrotizing Fasciitis
MeSH Terms: conditions — Fasciitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients and their significant others: Patients affected by necrotizing fasciitis and their significant others

SUMMARY:
Severe necrotizing soft tissue infection (NSTI), including necrotizing fasciitis, is a life threatening infection that spreads quickly to cutis, sub-cutis, fasciae and muscles. Approximately 40% of all patients with infections caused by S. Pyogenes develop a streptococcal toxic-shock syndrome. In these cases the mortality rates exceed 40% in spite of adequate treatment with antimicrobials. Due to the rapid progress, the extensive damage on soft tissues and high risk of death, the microbes are called "flesh-eating bacteria". The present study is a spin-off of the larger EU funded INFECT study, looking at the experiences of patient and family to understand the impact on every day life. The present prospective mixed methods study has the potential to provide important knowledge regarding the occurrence of early signs and symptoms of NSTI, quality of life 6 and 24 months after diagnosis, and how the care and treatment can be optimized and organized in a person/patient and family centered way. The study also aims at validate the SF 36 questionnaire for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with necrotizing fasciitis and their significant others
* Age above 18 yrs

Exclusion Criteria:

* Persons with dementia or severe psychiatric illness
* Persons that do not master the Scandinavian language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for necrotizing fasciitis at the three study sites
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 6 months
  Quantitative - health related quality of life Qualitative - patient experience
Quality of life | 24 months
  Quantitative - health related quality of life Qualitative - patient experience

SECONDARY OUTCOMES:
Quality of life of significant others | 6 months
  Quantitative - health related quality of life Qualitative - experience of significant others
Quality of life of significant others | 24 months
  Quantitative - health related quality of life Qualitative - experience of significant others

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Egron Thörn, MD, ass prof, Study Director — Sahlgrenska University Hospital
Locations (3):
- Rigshospitalet, Copenhagen, Denmark
- Sweden (2):
  - Sahlgrenska University hospital, Gothenburg
  - Karolinska Universitetssjukhuset, Solna